CLINICAL TRIAL: NCT06163820
Title: Bevacizumab and Immune chEckpoint Inhibitors Plus Hypofractionated Stereotactic radioTherapy for the Treatment of sympTomatic mElanoma bRain Metastases.
Brief Title: Bevacizumab and ICIs + hSRT in Symptomatic Melanoma Brain Metastases
Acronym: BETTER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05.21 BETTER
Record Dates: First submitted 2023-10-17; First posted 2023-12-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Melanoma Brain Metastases
MeSH Terms: interventions — Bevacizumab; Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: The trial is a phase I/II, single arm, unblinded, multi-centre dose de-escalation trial to evaluate the safety and efficacy of the combination of bevacizumab, with ipilimumab plus nivolumab, and hypofractionated stereotactic radiotherapy (hSRT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will receive the following:
  1. Bevacizumab 7.5 mg/kg every 3 weeks for 4 cycles
  2. Nivolumab 1 mg /kg + ipilimumab 3 mg/kg every 3 weeks for 4 cycles (induction phase) followed by nivolumab monotherapy at 480mg every 4 weeks (maintenance phase)
  3. hSRT (24-27Gy/3# or 25-30Gy/5#)
  Interventions: Drug: Bevacizumab; Drug: Ipilimumab; Drug: Nivolumab; Radiation: Hypofractionated stereotactic radiotherapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is a humanised monoclonal antibody with molecular weight 167kD that inhibits all isoforms of the vascular endothelial growth factor (VEGF) and is produced from a Chinese hamster ovary mammalian system. It has high specificity for isoform-A and has a half-life of ~21 days.
  Other Names: Avastin
Drug: Ipilimumab — Ipilimumab is an immune checkpoint inhibitor (ICI) that targets anti-tumour immunity. Ipilimumab is a recombinant human immunoglobulin monoclonal antibody that binds CTLA4 and blocks the interaction between CD80/86 and CTLA4.
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab ia an immune checkpoint inhibitor (ICI) that targets anti-tumour immunity. Nivolumab is a fully human monoclonal IgG4 antibody targeting PD-1 which demonstrates activity across a range of tumours.
  Other Names: Opdivo
Radiation: Hypofractionated stereotactic radiotherapy — Hypofractionated stereotactic radiotherapy (hSRT) will be delivered to previously untreated brain metastases in eligible participants. hSRT will be delivered to all symptomatic brain metastases, all brain metastases >1 cm and all brain metastases located in eloquent areas of the brain. hSRT will be commenced after the first cycle of nivolumab plus ipilimumab and completed before the second cycle of nivolumab plus ipilimumab. hSRT should be commenced within 1 week from the planning MRI.

SUMMARY:
Single arm phase I/II trial to evaluate the safety and efficacy of the combination of bevacizumab, with ipilimumab plus nivolumab, and hypofractionated stereotactic radiotherapy (hSRT) in patients with symptomatic melanoma brain metastases (MBM).

DETAILED DESCRIPTION:
Despite significantly improved clinical outcomes for patients with metastatic melanoma, the subset of patients with symptomatic MBM still fare poorly with treatment. The current standard of care for this group of patients is combined immune checkpoint blockade with ipilimumab and nivolumab, with local treatment with neurosurgery or stereotactic radiotherapy added for larger/more symptomatic lesions.

Bevacizumab has demonstrated evidence in the treatment of cerebral radiation necrosis and in a case series, promising symptomatic benefit in this group of patients. With strong empirical evidence of the ability to wean patients from steroids, mechanistically, bevacizumab may augment anti-tumour immunity from immune checkpoint blockade.

Bevacizumab will be administered 7 days prior to combination immunotherapy with ipilimumab and nivolumab and then given 28 days later to coincide with the second cycle of ipilimumab and nivolumab and thereafter every 3 weeks. The starting dose will be 7.5mg/kg, given intravenously, for a total of four cycles, and is consistent with the existing literature on the treatment of cerebral radiation necrosis.

This trial aims to determine the safety of bevacizumab, in combination with ipilimumab, nivolumab and hSRT, defined as no more than 1/6 patients experiencing a bevacizumab-related SAE in the initial phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically (or cytologically) proven metastatic melanoma, with radiologically confirmed brain metastases.
* 2. Symptomatic from brain metastases at the time of study enrolment, or brain metastases that requires corticosteroids for the management of neurological symptoms.
* 3. Intracranial lesions amenable to hypofractionated stereotactic radiotherapy. These are defined as all intracranial melanoma lesions greater or equal to 5 mm in diameter, all intracranial lesions that are causing symptoms, and all intracranial lesions located in the eloquent areas of the brain.
* 4. World Health Organisation (WHO) performance status of 0 - 2
* 5. At least one brain metastasis has to be symptomatic.
* 6. Laboratory tests required: Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1 x 109/L Platelet count ≥ 100 x 109/L Either: Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (Patients with isolated hyperbilirubinaemia due to Gilbert's syndrome are allowed.) Or: Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible Creatinine clearance ≥ 40 mL/min (Cockcroft-Gault or MDRD are acceptable)
* 7. Age ≥ 18 years
* 8. Able to provide informed written consent (signed and dated), attend trial site for study visits and be capable of co-operating with treatment and follow-up

Exclusion Criteria:

* 1. Prior radiotherapy to the brain
* 2. Active concurrent malignancy requiring systemic anti-cancer therapy within the last 2 years. Patients with any malignancy treated with curative intent and no evidence of disease will be eligible for this trial.
* 3. Prior systemic therapy for melanoma, unless given in the neoadjuvant or adjuvant setting for extracranial disease only, completed more than >6 months prior to enrolment in this trial and if administered with radiological proof of the absence of brain metastases
* 4. Inability to undergo MRI of the brain
* 5. Definitive leptomeningeal disease. Patients with equivocal leptomeningeal disease may be included on the trial after discussion with CPI.
* 6. Female patients who are pregnant or lactating. Patients who are able to become pregnant, must return a negative serum or urine pregnancy test before enrolment and agree to use two forms of contraception (one effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence, effective from signing the consent form, throughout the trial and for six months after any treatment for melanoma, radiotherapy or immunotherapy, are considered eligible.
* 7. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception or to sexual abstinence effective from the first administration of bevacizumab, throughout the trial and for six months afterwards after treatment the end-of-trial visit. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Men with pregnant or lactating partners must be advised to use barrier method contraception to prevent exposure of the foetus or neonate. Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* 8. Haemorrhage encompassing >50% of any lesion that is >10 mm in diameter (excluding surrounding oedema). A modern susceptibility-sensitive MRI sequence such as SWI is mandatory.
* 9. Brain metastases greater than 5 cm in maximal diameter
* 10. Increasing corticosteroid dose for 48 hours prior to initiation of study therapy OR current dexamethasone-equivalent dose of >8 mg per day
* 11. Major thoracic or abdominal surgery within 28 days prior to initiation of trial treatment
* 12. Neurosurgery within 14 days prior to initiation of trial treatment
* 13. Active or history of severe auto-immune disease requiring systemic anti-inflammatory therapy. Patients with well-controlled auto-immune diseases not requiring systemic anti-inflammatory therapy may be included after consultation with the CPI. Severe auto-immune respiratory disease will be excluded from the trial.
* 14. History of inflammatory bowel disease
* 15. Requirement for ongoing concurrent systemic immunosuppressive therapy (other than corticosteroids).
* 16. History of intra-abdominal inflammatory process within 6 months prior to initiation of trial treatment, including but not limited to peptic ulcer disease, diverticular disease or colitis.
* 17. History of abdominal or trachea-oesophageal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to initiation of trial treatment
* 18. History of intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition or tube feeding within 6 months prior to initiation of trial treatment
* 19. Any Grade ≥3 haemorrhage or bleeding event within 28 days of trial treatment initiation. Patients presenting with haemorrhagic brain metastases that have been adequately treated with neurosurgery are not excluded under this criterion but remain subject to criterion 12 pertaining to timing of neurosurgery.
* 20. Current use of full-dose anticoagulation or thrombolytic therapy within 10 days of initiation of trial treatment
* 21. Evidence of bleeding diatheses or significant coagulopathy
* 22. History of inadequately controlled arterial hypertension (systolic BP ≥160 mm Hg or diastolic BP ≥100 mm Hg despite maximal medical therapy); prior history of hypertensive crises or hypertensive encephalopathy
* 23. Concurrent congestive heart failure, prior history of NYHA class III/ IV cardiac disease, prior history of cardiac ischaemia or prior history of cardiac arrhythmia
* 24. Concurrent participation in another interventional clinical trial or intention to do so. Concurrent participation in an observational trial is acceptable.
* 25. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of bevacizumab, in combination with ipilimumab, nivolumab and hSRT | 5 years
  Number of participants with bevacizumab-related SAEs. A dose-limiting toxicity rate of <33% with a minimum of 3 patients treated will be considered safe.

SECONDARY OUTCOMES:
Determining the magnitude in reduction in prednisolone equivalent dose (relative to baseline dose) | 2 years
  The combination of a strict patient diary of corticosteroid dose, volumetric analysis of oedema on paired MRI samples with Peripheral blood mononuclear cells (PBMCs) to delineate immune cell subsets will allow proof-of-mechanism to be demonstrated.
  Specifically, if the proposed combination demonstrates preliminary activity, we will be able to demonstrate that this activity corresponds to a decrease in steroid dose (diary) which is permissible due to reduced oedema (volumetric analysis), resulting in augmented antitumour immunity (as evidence by increased peripheral antitumour immune cells). Finally, the inclusion of a health-related quality of life (QoL) analysis in this early phase clinical trial, may demonstrate that the reduction in steroid dose is clinically meaningful to patients.
Intracranial clinical benefit | 5 years
  The rate of intracranial clinical benefit, defined as the percentage of patients who had stable disease for at least 6 months after the initiation of treatment, complete response (CR), or partial response (PR)
Response rate | 5 years
  The rate of overall response (defined as the rate of complete or partial response)
Progression-free survival | 5 years
  The rate of intracranial, extracranial (systemic), and global progression-free survival (PFS)
Overall survival | 5 years
  Overall survival
Volume of vasogenic oedema | 2 years
  Determining the magnitude in reduction of the volume of vasogenic oedema around the brain metastases on MRI scan, after the administration of bevacizumab
To assess the patient-rated quality of life by the mean change from baseline quality of life scores [QLQ-C30] to the time of response, stable disease or progression. | 2 years
  We will assess utility-based health-related quality of life (HRQoL) of the combination of bevacizumab, with ipilimumab plus nivolumab, and hSRT using scores from the EORTC QLQ-C30 instrument transformed to QLU-C10D algorithm at baseline and 6-weekly for 6 months, then 12 weekly thereafter to identify resultant improvements in patients' QoL. In addition, the utility indices will be used to estimate quality-adjusted life years (QALYs).

OTHER OUTCOMES:
To correlate anti-tumour activity with the detection of putative biomarkers of response/resistance in paired blood samples. | 5 years
  Disease is measured according to the RECIST criteria (version 1.1). Imaging-based evaluation is preferred to evaluation by clinical examination when both methods have been used to assess the anti-tumour effect of a treatment. Overall response rate will be correlated to putative biomarkers.
Rate of cerebral radiation necrosis | 2 years
  To assess the impact of upfront bevacizumab on rates of cerebral radiation necrosis compared to historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Malaka Ameratunga, Study Chair — Monash University
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No